CLINICAL TRIAL: NCT04049630
Title: Randomized Clinical Trial, Double-blind, Dose-escalating of Drug Intensities, Evaluating the Safety and Efficacy of Levamisole in Loa Loa Microfilaremic Patients
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of Levamisole in Loa Loa Microfilaremic Patients
Acronym: EOLoa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Programme National de Lutte contre l'Onchocercose, Republic of the Congo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EOLoa/LEV
Record Dates: First submitted 2019-07-26; First posted 2019-08-08 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Onchocerciasis, Ocular; Loiasis
MeSH Terms: conditions — Onchocerciasis, Ocular; Loiasis | interventions — Levamisole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LEV 1 mg/kg (Experimental): Tablets of LEV at 1 mg/kg will be administrated to the participant ; in single dose only one time. The number of tablets of LEV of 50 mg or 10 mg will be adapted according to the weight of the participant.
  Interventions: Drug: LEV 1 mg/kg; Drug: Placebo
- LEV 1,5 mg/kg (Experimental): Tablet of LEV at 1,5 mg/kg will be administrated to the participant ; in single dose only one time. The number of tablets of LEV of 50 mg or 10 mg will be adapted according to the weight of the participant.
  Interventions: Drug: LEV 1,5 mg/kg; Drug: Placebo
- LEV 2,5 mg/kg (Experimental): Tablet of LEV at 2,5 mg/kg will be administrated to the participant ; in single dose only one time. The number of tablets of LEV of 50 mg or 10 mg will be adapted according to the weight of the participant.
  Interventions: Drug: LEV 2,5 mg/kg; Drug: Placebo
- Placebo (Placebo Comparator): Tablets of placebo will be administrated to the participant in single dose only one time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEV 1 mg/kg — A combinaison of LEV 10 mg, 50 mg, and placebo will be adapted to the weight ; all the tablets will be blinded, and each participant will receive 5 tablets.
  Arms: LEV 1 mg/kg
Drug: LEV 1,5 mg/kg — A combinaison of LEV 10 mg, 50 mg, and placebo will be adapted to the weight ; all the tablets will be blinded, and each participant will receive 5 tablets.
  Arms: LEV 1,5 mg/kg
Drug: LEV 2,5 mg/kg — A combinaison of LEV 10 mg, 50 mg, and placebo will be adapted to the weight ; all the tablets will be blinded, and each participant will receive 5 tablets.
  Arms: LEV 2,5 mg/kg
Drug: Placebo — 5 tablets of placebo will be administrated to the participants.

SUMMARY:
This study aims at evaluating the safety and efficacy of levamisole in patients with loiasis infection.

DETAILED DESCRIPTION:
This clinical trial will be conducted in Republic of Congo. This is a pragmatic and adaptative randomized, double-blind clinical trial. Levamisole will be tested at 1 and 1,5 mg/kg, and compared to placebo (36:36:36); or 2,5 mg/kg compared to placebo (36:36) in case of adaptation of the dose for cohorts II and III.

We will perform three cohorts of patients according to the microfilarial density : 1-1,999 mf/ml, 1-14,999 mf/ml, and all microfilaremic individuals; in order to respect the safety potentially related to loiasis.

The first cohort was to evaluate the most appropriate dose of levamisole, with a possibility to increase (to 2.5 mg/kg) the dose of levamisole for the cohorts II and III in case of lack of efficacy and in case of good safety profil.

ELIGIBILITY:
Inclusion Criteria:

* Written consent written, signed (or with thumbprint) and dated
* Aged 18 to 65 inclusive
* Individual microfilarial density ≥ 1mf/mL
* Body weight ≥ 40 kg in women and ≥ 45 kg in men; and less than 85 kg
* In good health condition, as determined by the medical questionnaire and the general clinical examination: absence of acute or chronic infection

Exclusion Criteria:

* Participation in any study other than purely observational, in the 4 weeks preceding this study (determined by the theoretical date of administration of LEV or placebo).
* Any vaccination in the 4 weeks preceding this study.
* Acute infection requiring a treatment in the 10 days preceding this study, determined by the anamnesis during the medical interview (example: pulmonary infection, ENT, digestive, cutaneous, with implementation of an antibiotic treatment or not)
* Warfarin treatment
* Treatment with clozapine, phenythiazines, sulfasalazine, carbamazepine, synthetic antithyroid, ticlopidine, cimetidine, and gold salts: whether it is a long-term treatment, or a treatment given in a single dose 10 days before the start of treatment for the clinical trial (precaution of use compared to the risk of agranulocytosis of immuno-allergic or toxic origin)
* Known immunosuppressive pathology
* Past or current history of neurological (including epilepsy) or neuropsychiatric disease
* History of agranulocytosis
* Consumption of alcohol, taking cocaine or other drugs of abuse in the 72 hours preceding the administration of the treatment of the test determined by the anamnesis during the medical interview
* Any condition, in the opinion of the investigator, which exposes the subject to an undue risk
* Known intolerance to levamisole
* Subjects who gave blood in the 8 weeks before entry into the study, with a standard volume (> 500 mL)
* During the clinical examination: symptoms, physical signs or biological constants suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, cutaneous, immunodeficiency, psychiatric disorders and other abnormalities likely to interfere with the interpretation results of the test. The doctor may then give a favorable or unfavorable opinion for the inclusion of the participant
* Taking IVM and / or LEV during the last six months; and / or mebendazole or albendazole in the last month
* Pregnant and lactating women (based on self-declaration)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of levamisole | 1 week
  Absence of severe adverse events during the first week
Incidence of adverse events with levamisole | 1 week
  Proportion of adverse events during the first week

SECONDARY OUTCOMES:
Efficacy of levamisole | Day 2, Day 7, and Month 1
  Proportion of reduction of the microfilarial density of Loa loa at Day 2, Day 7, and Month 1
Proportion of individuals without microfilariae of Loa loa | Day 7 and 1 Month
  Proportion of individuals with a diminution of 40% and 80% and more of the microfilarial density at Day 7 and Month 1

CONTACTS AND LOCATIONS:
Locations (1):
- Secteur opérationnelle de la Santé, Ministère de la Santé et de la Population, Sibiti, Republic of the Congo

REFERENCES:
- [Derived] Campillo JT, Bikita P, Hemilembolo M, Louya F, Missamou F, Pion SDS, Boussinesq M, Chesnais C. Safety and Efficacy of Levamisole in Loiasis: A Randomized, Placebo-controlled, Double-blind Clinical Trial. Clin Infect Dis. 2022 Aug 24;75(1):19-27. doi: 10.1093/cid/ciab906. PMID 34651190